CLINICAL TRIAL: NCT01446107
Title: A Randomized Controlled Trial on the Effectiveness of Fissure Sealant and Topical Fluoride Application in Preventing Dental Caries
Brief Title: Effectiveness of Fissure Sealant and Topical Fluoride Application in Preventing Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW06-402T/1427
Record Dates: First submitted 2011-09-23; First posted 2011-10-05 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2011-09

CONDITIONS: Dental Caries
Keywords: tooth decay; fluoride; sealant; prevention
MeSH Terms: conditions — Dental Caries | interventions — silver fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fissure sealant (Experimental): single placement of resin fissure sealant on tooth surface
  Interventions: Other: placement of fissure sealant
- fluoride varnish (Experimental): application of a 5% sodium fluoride varnish every 6 months
  Interventions: Other: fluoride varnish
- SDF solution (Experimental): application of a 38% silver diamine fluoride solution onto tooth surface every year
  Interventions: Other: silver fluoride
- control (Placebo Comparator): application of water onto tooth surface every year
  Interventions: Other: placebo control

INTERVENTIONS:
Other: placement of fissure sealant — placement of resin-based fissure sealant at baseline without replacement
  Arms: fissure sealant
Other: fluoride varnish — topical applications of a 5% sodium fluoride (NaF) varnish onto tooth surface every 6 months
  Arms: fluoride varnish
Other: silver fluoride — topical applications of a 38% silver diamine fluoride (SDF) solution onto tooth surface every year
  Arms: SDF solution
Other: placebo control — application of water onto tooth surface every year
  Arms: control

SUMMARY:
Nearly half of the 12-year-old children in China have dental caries (tooth decay) and most of the lesions are in the fissures of the first permanent molars. This study aims to investigate the effectiveness of three methods in preventing fissure caries in permanent teeth in Chinese children, namely resin fissure sealant, sodium fluoride varnish, and silver diamine fluoride solution. The cost-effectiveness of these methods will also be compared. About 400 children, aged 8 to 9 years, will be recruited. Clinical examination of the children will be conducted in school using portable dental lights and instruments to identify teeth that need caries prevention. The children will be randomly allocated to one of the three test or the control groups. Treatments will be provided in the study primary schools according to standard clinical protocols. Follow-up examinations will be carried out every six months for 30 months to assess whether the preventive methods are successful, i.e. no dental caries develops in the treated teeth. The findings of this study will be of great value to dentists and public health authorities in deciding on the most appropriate dental caries prevention programme for school children in China and other developing countries.

ELIGIBILITY:
Inclusion Criteria:

* school children in good general health
* have at least one permanent first molars that has deep occlusal fissures, or fissures with signs of early caries

Exclusion Criteria:

* children with major systemic disease or taking long-term medications
* not cooperative or refuse dental treatments

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
dental caries | 3 years
  tooth decay appearing as a cavity on tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Edward CM Lo, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Liu BY, Lo EC, Chu CH, Lin HC. Randomized trial on fluorides and sealants for fissure caries prevention. J Dent Res. 2012 Aug;91(8):753-8. doi: 10.1177/0022034512452278. Epub 2012 Jun 26. PMID 22736448